CLINICAL TRIAL: NCT02396576
Title: Using Telehealth to Deliver Mental Health Services in Primary Care Settings for Children in Underserved Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Tumaini R Coker, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IH-12-11-4168
Record Dates: First submitted 2015-03-04; First posted 2015-03-24 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Developmental, Behavioral and Mental Health; Adhd; Depression; Anxiety; Developmental Delay; Autism; Behavioral Problems
MeSH Terms: conditions — Behavior; Psychological Well-Being; Attention Deficit Disorder with Hyperactivity; Depression; Anxiety Disorders; Learning Disabilities; Autistic Disorder; Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): NEVHC has two main Department of Mental Health (DMH) contracted clinical partners where the majority of the patients are referred to -these are Child and Family Guidance Center (CFGC) in the San Fernando Valley and Child and Family Center (CFC) in the Santa Clarita Valley.
- Telehealth Intervention (Experimental): The telehealth model will enhance patient coordination as well as clinician communication via live videoconferencing. Developmental behavioral services will be provided by a Developmental Behavioral Pediatrician (DBP) housed at UCLA from Children's Hospital Los Angeles (CHLA). Mental Health services will be provided by Child Family Center (CFC) and Child Family Guidance Center (CFGC). The location of the telehealth visit will be at the same clinic location as the index PCP visit with a telehealth coordinator facilitating the encounter between patient and clinicians.The clinician communication will be enhanced through monthly telehealth topic-based educational sessions as well as case-based educational sessions for the transfer cases.
  Interventions: Behavioral: Telehealth Intervention

INTERVENTIONS:
Behavioral: Telehealth Intervention — The telehealth model will integrate developmental, behavioral, (DB) and mental health services (MH) into pediatric primary care using videoconferencing that will be tested with children in low-income, urban communities.
  Arms: Telehealth Intervention

SUMMARY:
In partnership with a multi-site, Los Angeles-area community clinic consortium, North East Valley Health Corporation (NEVHC), the investigators will use telehealth to integrate pediatric developmental, behavioral and mental health (DB/MH) services into primary care for low-income, publicly insured children. During Project Year 1, the investigators used qualitative methods to conduct and analyze interviews with parents, clinicians, and staff at NEVHC to assess their perspectives on the delivery of child DB/MH services and on a potential telehealth-based patient visit, coordination, and clinician education system for the provision of DB/MH specialty care in primary care settings to children ages 5-12. This data was used in a stakeholder-engaged process to customize a telehealth-based delivery system for pediatric DB/MH services that can be integrated into primary care settings.

During Project Years 2-3, the investigators will conduct a cluster randomized controlled trial (RCT) to compare the customized telehealth-based patient visit, coordination, and clinician education system to the usual in-person, community- based referral system at NEVHC. This study will examine whether a telehealth developmental, behavioral and mental health delivery model can be an effective, efficient, and family-centered way to provide integrated DB/MH services to children in low-income communities.

DETAILED DESCRIPTION:
There are three main parts to the basic template of this telehealth intervention:

1. Real-time videoconference patient visits. Patients who need a specialty visit with a developmental/behavioral pediatrician will be scheduled for a telehealth visit (with the patient at the primary care clinical site and the subspecialists located at a University of California, Los Angeles (UCLA) telehealth site). Patients who need a psych/MH referral will initially connect with the mental health clinic (MHC) via telehealth. Therapy visits and the initial psychiatric assessment for medications are in person. Follow up psychiatric visits are via telehealth.
2. Enhanced clinician communication and patient coordination. Providers will use telehealth capabilities to communicate with each other about patient care and coordination issues, including diagnostic decisions, management strategies, and other patient care coordination activities.
3. Clinical educational sessions for clinicians. The telehealth equipment will also be used for real-time videoconference educational sessions to help primary care clinicians and specialty care clinicians share knowledge and experience that can translate into greater improvements for patient care.

The investigators will compare the new customized telehealth-based patient visit, coordination, and clinician education system to the usual in-person, community based referral system at NEVHC. Patients scheduled for a telehealth visit will receive a phone reminder 2 days before the visit. The location of the telehealth visit will be at the same clinic location as the index primary care provider (PCP) visit. Upon arrival for their telehealth visit, parents will be sent to a typical patient encounter room at the clinical site. The room will be set up for a telehealth visit with telehealth equipment, two chairs for the parent(s) and a small table with chairs and toys for the child and any siblings that arrive with the family. The camera will be set up to allow the specialty provider to have full view of the examination room. The system uses a multifunctional camera with zoom and pan (side to side) capabilities; the investigators will utilize a high-speed internet connection at NEVHC for optimal connection speed.

A bilingual (Spanish and English) telehealth coordinator will greet the parents and coordinate the visit at the NEVHC end. The telehealth coordinator is present at the NEVHC end of the telehealth visit for the duration of the visit. The telehealth coordinator ensures that the camera and microphones are operating correctly, positions the camera as necessary, conducts a volume and vision check, and as the exam proceeds, provides Spanish language interpretation if necessary.

The clinical encounter proceeds as a typical "in-person" encounter.

The developmental behavioral services in the telehealth-based patient visit will be provided by a developmental behavioral pediatrician (DBP) housed at UCLA from Children's Hospital Los Angeles (CHLA). The telehealth coordinator will call parent to inform parents of their DBP appointment date/time and will explain the telehealth visit.

The mental health services will be performed by psychiatrists at CFGC and CFC. The telehealth specialty physician will conduct the typical history, review of information brought by the parent to the visit, focused behavioral observations, and a general visual inspection, with assistance from the telehealth coordinator on the distal end. At the end of the visit, the telehealth coordinator will assist the physician in setting up any follow-up plans with the family. The telehealth coordinator will then prepare for the next scheduled patient.

The other two components of the telehealth system include clinical educational sessions and clinician communication and patient coordination sessions. As part of our ongoing stakeholder engagement process, the investigators will hold a telehealth primary care-mental health educational session via videoconference monthly. These sessions are topic-based webinars and case-based educational sessions for the transfer cases. Sessions will alternate between webinars and case-based educational sessions. The session will include the child psychiatrist(s), and the NEVHC PCPs; each session will be held during the clinic's lunch hour for about 45 minutes, based on the NEVHC PCP availability. There will be 9 topic-based webinar sessions during the intervention period. The first 4 sessions will focus on referral indications and recommendations for the most common child MH symptoms. Topics include: guidelines for referral to CFGC/CFC (e.g., when not to refer), diagnosis and management of attention deficit hyperactivity disorder, anxiety, and depression, and diagnostic criteria for Oppositional Defiant Disorder and PTSD. the investigators will also conduct some sessions on primary care topics (e.g., anorexia nervosa) for mental health providers.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian with child between the ages of 5 to 12
* Must speak English or Spanish
* Child has been referred by primary care doctor for mental health or developmental behavioral services

Exclusion Criteria:

* Parent /Guardian under 18 years of age
* Parent employed by Northeast Valley Health Corporation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Access to specialty services- Referral time | 6 month post-enrollment
  Referral process from baseline to 6 month post-enrollment. Parent reported time from initial referral to first specialty visit as reported by parents on 6 month post-enrollment survey.
Access to specialty services- Travel | 6 month post-enrollment
  Parent reported number of miles traveled and commute time to initial visit as reported by parents on 6 month post-enrollment survey.
Access to specialty services- Missed school/work | 6 month post enrollment
  Parent reported number of days missed from school/work as reported by parents on 6 month post-enrollment survey.
Access to specialty services- Out of pocket cost | 6 month post-enrollment
  Parent reported amount of money spent for daycare and specialty services as reported by parents on 6 month post-enrollment survey.
Access to specialty services- Visits | 6 month post-enrollment
  Number of specialty visits attended as reported by parents on 6 month post-enrollment survey.

SECONDARY OUTCOMES:
Quality of care measures | 6 month post-enrollment
  Parent reported quality of care measures as measured by the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Clinician and Group Survey. Three measures will be utilized from CAHPS; 1.Timely Appointment, Care and Information, 2. Providers Communication with Patients, and 3. Patients' Rating of Providers.
Child Behavior measures | 6 month post-enrollment
  Parent reported child behavior as measured by Pediatric Quality of Life (PedsQL), and Pediatric Symptom Checklist.
Provider coordination- Communication | 6 month post-enrollment
  Provider reported level of communication between PCP and specialists as measured by the communication measure from the California Mental Health Services Authority Integrated Behavior Health Care (IBHC).
Provider coordination- Comfort level | 6 month post-enrollment
  Provider reported comfort level of diagnosis, medication initiation, medication management, and patient monitoring as reported by providers on 6 month post-enrollment survey.

CONTACTS AND LOCATIONS:
Overall Officials: Tumaini Coker, MD, Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (6):
  - Northeast Valley Health Corporation- Canoga Park, Canoga Park, California
  - Northeast Valley Health Corporation- Pacoima, Pacoima, California
  - Northeast Valley Health Corporation- San Fernando, San Fernando, California
  - Northeast Valley Health Corporation- Santa Clarita, Santa Clarita, California
  - Northeast Valley Health Corporation- Valencia, Valencia, California
  - Northeast Valley Health Corporation- Van Nuys, Van Nuys, California

REFERENCES:
- [Derived] Coker TR, Porras-Javier L, Zhang L, Soares N, Park C, Patel A, Tang L, Chung PJ, Zima BT. A Telehealth-Enhanced Referral Process in Pediatric Primary Care: A Cluster Randomized Trial. Pediatrics. 2019 Mar;143(3):e20182738. doi: 10.1542/peds.2018-2738. Epub 2019 Feb 15. PMID 30770523